CLINICAL TRIAL: NCT07148999
Title: An Advanced Decision Support Tool for Personalized Medicine for IVF Using Modeling and Optimization for PPOS
Brief Title: An Advanced Decision Support Tool for Personalized Medicine for IVF Using Modeling and Optimization for Provera
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Urmila DIwekar (Industry)
Collaborators: IVF Academy of USA (Unknown); Positivf Fertility (Unknown)
Responsible Party: Sponsor-Investigator, Urmila DIwekar, President, Stochastic Research Technologies LLC
Organization: Stochastic Research Technologies LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPOS-1
Record Dates: First submitted 2025-08-15; First posted 2025-08-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Infertility (IVF Patients)
Keywords: Opt-IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: The primary protocol used in this trial is a progesterone-primed ovarian stimulation (PPOS).
  This is a multi-site cohort with two arms (one arm for the intervention and one arm for the traditional approach), a randomized clinical trial involving more than 100 patients. The clinical trial will be registered on ClinicalTrials.gov. It is a parallel trial with a 1:1 allocation. A Simple Randomization method will assign patients to the intervention and control groups using a lottery method. The generation of random sequences will be carried out by Dr. Diwekar, who will not be involved in the clinical administration of the trial. The patients will be registered and assigned to different groups separately at each center. The allocation will be masked until participants are ready to receive the intervention. An administrator, who will not be a clinical investigator, will allocate a participant to one arm using the random sequences generated prior to the trial. The clinicians, participants,
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): This arm will get dosage prescribed by the doctor
  Interventions: Other: Control
- Opt-IVF (Experimental): This arm patients will get dosage provided by Opt-IVF
  Interventions: Combination Product: Opt-IVF

INTERVENTIONS:
Combination Product: Opt-IVF — Opt-IVF provides optimized dosage profile for each patient
  Arms: Opt-IVF
Other: Control — Physicians will decide the dosage for each day for patients
  Arms: Control

SUMMARY:
A clinical trial will determine the effectiveness of using the Opt-IVF decision support tool for each patient's personalized and optimal drug dosage profile in the United States.

DETAILED DESCRIPTION:
This will be a two-arm randomized clinical trial involving more than 100 patients; one arm will undergo superovulation using dosages predicted by the decision support tool, while the other will undergo the current standard treatment. The research question is whether outcomes of patient dosage treatment using Opt-IVF are better or similar to the current practice. We will compare the outcomes of the two groups of patients in terms of the numbers and percentage of mature follicles retrieved at the end of each cycle, total FSH and HMG dosages used, and the number of required testing days for that cycle, total number of M2s, Number of embryos, Number of Grade A embryos and Number of Grade A blastocysts.

The trial is for research purposes only. The current tool has not been submitted for any regulatory body approval.

ELIGIBILITY:
Inclusion Criteria:

* infertile women

Exclusion Criteria:

All female patients who will not undergo IVF or whose cycles will be converted to IUI. Male patients will not be enrolled in this study. No donor cycles.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This treatment is for women undergoing IVF
Enrollment: 200 (Estimated)
Dates: Start 2025-09-23 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Total Gonadotropin Dosage | Two weeks after the start of the cycle
  Total Gonadotropin Dosage for the cycle
Total Oocytes Retrieved | Two weeks after the start of the stimulation cycle
  Total Oocytes Retrieved
M2 Oocytes | Two weeks after the start of the stimulation cycle
  Total M2 Oocytes
Total Embryos Formed | Two weeks after the start of stimulation cycle
  Total Embryos Formed
Grade A embryos/Blastocytes | Three weeks after the start of stimulation cycle
  Grade A Day 3 Embryos or Grade A Day 5 Blastocytes

SECONDARY OUTCOMES:
Pregnancy Rates | one month after first transfer
  Cycle pregnancy rate till the first transfer

CONTACTS AND LOCATIONS:
Overall Officials: Paul Magarelli, M.D., Ph.D., Principal Investigator — IVF Academy USA; Francesco Arredondo, MD, Ph.D., Study Director — Positivf Fertility
Locations (2):
- United States (2):
  - Positivf Fertility, Houston, Texas
  - Positivf Fertility, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will be available by contacting Dr. Urmila Diwekar
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the trial
Access Criteria: by contacting Dr. Diwekar

REFERENCES:
- [Background] Diwekar et al., A multicenter randomized clinical trial with a novel decision support tool to improve IVF success, Reproduction and Fertility, 6(3), e250004, 2025.DOI: https://doi.org/10.1530/RAF-25-0004
- [Background] Diwekar U, Gupta S, Gahlan A, Hota S, Murdia K, Murdia N, Chandra V, Bhoi N, Joag S. A new decision-support tool in a multi-center randomized trial for personalized, optimized, and simplified fertility treatment in non-PCOS patients. Reprod Fertil. 2024 Sep 16;5(3):e240013. doi: 10.1530/RAF-24-0013. Print 2024 Jul 1. PMID 39159260
- [Background] Nisal A, Diwekar U, Bhalerao V. Personalized medicine for in vitro fertilization procedure using modeling and optimal control. J Theor Biol. 2020 Feb 21;487:110105. doi: 10.1016/j.jtbi.2019.110105. Epub 2019 Dec 3. PMID 31809718
- See also: all clinical publications are available here — https://opt-ivf.com/studies.html